CLINICAL TRIAL: NCT05971784
Title: The Effect of Upper Extremity Telerehabilitation on Balance and Gait in Parkinson's Patients
Brief Title: The Effect of Upper Extremity Telerehabilitation on Balance and Gait
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Sefa Eldemir, Principal Investigator, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6- PD-Balance-Telereh-RCT
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Task oriented training; Balance; Gait
MeSH Terms: conditions — Parkinson Disease | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Two groups as exercise group and control group
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation group (Experimental): In addition to the exercise program consisting of balance and walking activities, the group will receive task-oriented upper extremity training via telerehabilitation accompanied by a physiotherapist.
  Interventions: Other: Telerehabilitation Group
- Control group (Experimental): The group that will receive a home exercise program consisting of only balance and walking activities
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Telerehabilitation Group — The group that will receive upper extremity training via telerehabilitation in addition to an exercise program consisting of balance and walking activities
  Arms: Telerehabilitation group
Other: Control Group — The group that will receive an exercise program consisting of balance and walking activities
  Arms: Control group

SUMMARY:
Parkinson's Disease (PD) is a disease that affects the upper extremity functional skills with clinical findings such as bradykinesia, rigidity, and hypokinesia and causes limitations in the daily living activities of the patients. The influence of fine dexterity, reaching, and grasping movements greatly affects the daily living activities of the patients. Medical treatment and surgical approaches are frequently used among the treatment options for PD today. Physiotherapy and rehabilitation approaches for progressive functional loss in PD, together with optimal medical and surgical treatment, form the basis of PD treatment. Recently, it has been stated that intensive and task-specific rehabilitation interventions in the field of physiotherapy and rehabilitation will be more effective than traditional rehabilitation approaches. On the other hand, telerehabilitation approaches, the use of which has increased rapidly due to technological developments in recent times, enables the delivery of rehabilitation services to patients in distant places by using communication technologies. For this purpose, it is highly valuable to implement a task-oriented training (TOT) program based on motor learning-based principles, which consists of intense exercise content, through telerehabilitation. Although there are very few studies investigating the effectiveness of telerehabilitation-based TOT in PD, these studies have shown that upper extremity motor performance, activities of daily living, and quality of life are improved. On the other hand, no study has been found showing the effect of upper extremity TOT applied through telerehabilitation on balance and walking. Therefore, there is a need to investigate the effectiveness of telerehabilitation-based TOT exercises on balance and walking.

DETAILED DESCRIPTION:
This study is a randomized controlled study. The patients will be randomly divided into two groups exercise and control. Balance and walking exercises consisting of 3 days a week for 6 weeks will be given to both groups as a home program. In addition, the exercise group will receive Task-oriented Training (TOT) based telerehabilitation via video conferencing 3 days a week for 6 weeks. TOT will be formed from daily life activities such as reaching out, grasping, writing, and manual skills, which are frequently used in daily life. As the outcome measures, disease severity, and disability, balance, and gait will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 40- 80 years of age
* Having diagnosed with "Parkinson's Disease" by a specialist physician
* Having between 1-3 stages according to the Hoehn and Yahr Scale
* Mini-Mental Test score more than or equal 24

Exclusion Criteria:

- Any orthopedic, vision, hearing, cardiovascular, or perception problems that may affect the research results

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Static Balance- Baseline | Assessment will be conducted before the intervention
  Assessment will be made with a Biodex Balance System
Static Balance- Post intervention | Assessment will be conducted immediately after the intervention
  Assessment will be made with a Biodex Balance System
Gait- Baseline | Assessment will be conducted before the intervention
  Assessment will be made with the Time up and Go Test
Gait- Post intervention | Assessment will be conducted immediately after the intervention
  Assessment will be made with the Time up and Go Test
Balance- Baseline | Assessment will be conducted before the intervention
  Assessment will be made with the Berg Balance Scale
Balance- Post intervention | Assessment will be conducted immediately after the intervention
  Assessment will be made with the Berg Balance Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Sivas Cumhuriyet University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data but when the statistical analysis of all data is made, all results will be shared.

REFERENCES:
- [Result] Eldemir S, Guclu-Gunduz A, Eldemir K, Saygili F, Yilmaz R, Akbostanci MC. The effect of task-oriented circuit training-based telerehabilitation on upper extremity motor functions in patients with Parkinson's disease: A randomized controlled trial. Parkinsonism Relat Disord. 2023 Apr;109:105334. doi: 10.1016/j.parkreldis.2023.105334. Epub 2023 Feb 28. PMID 36917914